CLINICAL TRIAL: NCT01786109
Title: Study on the Effect of Cannabinoid Agonist on Gastrointestinal and Colonic Motor and Sensory Functions in Patients With Diarrhea-Predominant Irritable Bowel Syndrome
Brief Title: Effect of a Cannabinoid Agonist on Colonic Sensory Functions in Patients With Irritable Bowel Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Camilleri (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor-Investigator, Michael Camilleri, Professor of Medicine, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 08-008314 Part B; R01DK079866 (NIH); UL1RR024150 (NIH)
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Results first posted 2013-03-13 (Estimated); Last update posted 2013-03-14 (Estimated); Status verified 2013-03

CONDITIONS: Irritable Bowel Syndrome
Keywords: anandamide; cannabinoid; fatty acid amide hydrolase; gastric; motility; small bowel; sensory; motor
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Dronabinol 2.5 mg (Experimental): One dose of dronabinol 2.5 mg was taken orally with water.
  Interventions: Drug: Dronabinol
- Dronabinol 5 mg (Experimental): One dose of dronabinol 5 mg was taken orally with water.
  Interventions: Drug: Dronabinol
- Placebo (Placebo Comparator): One dose of placebo was taken orally with water.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol — Dronabinol is a synthetic delta-9-tetrahydrocannabinol, a nonselective cannabinoid agonist. Subjects received one dose of either 2.5 mg or 5 mg orally with water.
  Other Names: Marimol
  Arms: Dronabinol 2.5 mg; Dronabinol 5 mg
Drug: Placebo — Placebo will match study drug; taken as one dose orally with water.
  Arms: Placebo

SUMMARY:
Irritable bowel syndrome (IBS) affects about 15% of the U.S. population. There are still no effective and safe medications approved for the treatment of abdominal pain associated with bowel symptoms in IBS. This study will investigate the effects of an approved medication, Dronabinol, on the movement of food through the stomach and colon in subjects with a history of diarrhea-predominant Irritable Bowel Syndrome (D-IBS).

DETAILED DESCRIPTION:
Irritable bowel syndrome (IBS) affects about 15% of the U.S. population. Despite increasing understanding of the pathophysiology of IBS, there is no effective medication approved for the treatment of abdominal pain associated with IBS. Cannabinoid receptors (CBR) are on cholinergic neurons in the brain stem, stomach and colon. A cannabinoid receptor 1 (CB1) antagonist, rimonabant, is effective in induction of weight loss; however, the mechanism of this benefit is unclear. Human studies from this lab show that a CBR agonist, dronabinol, inhibits gastric and colonic motility, which may alter appetite or satiation in obesity, and may have potential in the treatment of IBS. The overall focus of the study is on the mechanisms involved in the modulation of gastric and colonic motor and sensory functions by cannabinoid receptors (CBR) in health and in IBS. CB1 receptors are also involved in nociception and in mediating inflammation which are increasingly recognized as being potential pathophysiological mechanisms in IBS.

All participants underwent the following procedures:

1. Documentation of eligibility, screening questionnaires and physical examination, including exclusion of rectal evacuation disorder by standard clinical evaluation within the past 12 months; this was important to ensure the diarrhea was not secondary to "retention with overflow".
2. Bowel preparation with PEG and electrolyte-containing oral colonic lavage solution, followed by a 12 hour fast.
3. Colonic testing of compliance, tone, motility and sensation measurement. Colonic compliance, fasting tone, sensory thresholds and sensory ratings in response to random-order phasic distensions were performed before treatment was administered. Then medication was ingested, and after 60 minutes, the same studies were performed that is compliance, fasting tone, sensory thresholds and sensory ratings in response to random-order phasic distensions. Participants also filled in responses to questionnaires (using 100 mm VAS scales) to describe their sense of tiredness, peace, worry and activity at the time of the measurements of sensation. Finally, participants ingested a standard chocolate 1000 kcal milkshake meal, and postprandial colonic tone and motility were measured for one hour.
4. With appropriate consent, a venous blood sample was obtained from each participant for DNA extraction; this will be used in ongoing pharmacogenomics studies.

Note: This study is related to NCT01253408, part A of the same protocol. Part A explored the effect of dronabinol on gastric and colonic motor functions.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years
* Positive for IBS symptoms by Rome III criteria
* No prior abdominal surgery (except appendectomy or cholecystectomy
* Score of 10 or less on either Anxiety or Depression on the Hospital Anxiety/Depression Inventory

Exclusion Criteria:

* Patients with significant depression (score of greater than 10 on Hospital Depression Inventory
* Patients with anxiety (score of greater than 10 on Hospital Anxiety Inventory. However, patients on stable doses of selective serotonin inhibitors (SSRIs) or low dose of tricyclic antidepressants will be eligible.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2009-09; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Camilleri, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Background] Wong BS, Camilleri M, Eckert D, Carlson P, Ryks M, Burton D, Zinsmeister AR. Randomized pharmacodynamic and pharmacogenetic trial of dronabinol effects on colon transit in irritable bowel syndrome-diarrhea. Neurogastroenterol Motil. 2012 Apr;24(4):358-e169. doi: 10.1111/j.1365-2982.2011.01874.x. Epub 2012 Jan 30. PMID 22288893
- [Result] Wong BS, Camilleri M, Busciglio I, Carlson P, Szarka LA, Burton D, Zinsmeister AR. Pharmacogenetic trial of a cannabinoid agonist shows reduced fasting colonic motility in patients with nonconstipated irritable bowel syndrome. Gastroenterology. 2011 Nov;141(5):1638-47.e1-7. doi: 10.1053/j.gastro.2011.07.036. Epub 2011 Jul 29. PMID 21803011
- See also: Link to Part A of this study, results for GI and colonic motor functions, n=36 — http://clinicaltrials.gov/show/NCT01253408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All participants were recruited from a database of patients with irritable bowel syndrome (IBS) who reside within 120 miles of Rochester, Minnesota
Groups:
- Dronabinol 2.5 mg: One dose of dronabinol 2.5 mg will be taken orally with water.
- Dronabinol 5 mg: One dose of dronabinol 5 mg will be taken orally with water.
- Placebo: One dose of placebo will be taken orally with water.
Period: Overall Study
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Started | 24 | 24 | 27
Completed | 23 | 24 | 25
Not Completed | 1 | 0 | 2
Not completed — fail manometry barostat tube placement | 1 | 0 | 0
Not completed — unrelated illness | 0 | 0 | 1
Not completed — adverse effects colon preparation | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo | Total
Number analyzed (Participants) | 24 | 24 | 27 | 75
Age Continuous [Mean (Standard Deviation); unit: years] | 36.1 (2.5) | 43.7 (2.1) | 43.2 (2.5) | 40.8 (11.935)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 23 | 24 | 69
  Male | 2 | 1 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 24 | 24 | 27 | 75
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 26.7 (1.0) | 29.7 (1.1) | 28.9 (1.2) | 28.3 (5.5)

OUTCOME MEASURES:

1. Primary Outcome: Colonic Compliance at Pressure at Half-Maximum Volume (Pr 1/2)
Description: Colonic compliance is a measure of the "stiffness" of the colon, that is, what pressure was needed to reach half the maximum volume of the colon.
  After the barostat catheter was inserted in the colon, the catheter was connected to a barostat machine. After an initial conditioning distension to 20 mm Hg, colonic compliance was measured by step-wise inflation with increments of 4 mm Hg up to 64 mm Hg. Colonic compliance was analyzed by a validated linear interpolation method. The pressure at half maximum volume serves as a summary of colonic compliance.
Time Frame: 1 hour after drug was ingested
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: mL/mm Hg
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
mL/mm Hg | 17.57 (0.935) | 16.2 (1.03) | 18.76 (1.13)

2. Secondary Outcome: Postprandial Change in Colonic Tone
Description: Colonic tone is a measurement of the volume of the colon. Colonic tone was assessed by noting the changes in the balloon volume in the presence of a constant operating pressure in the balloon (in the barostat-manometric assembly placed in the colon.)
Time Frame: 1 hour after ingestion of standard meal
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: mL
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
mL | 30.34 (4.76) | 27.41 (3.35) | 26.31 (4.81)

3. Secondary Outcome: Post-treatment Sensory Threshold for First Perception of Pain
Description: The sensory threshold for first perception of pain was measured by stepwise inflation in increments of 4 mm Hg at 60 second intervals up to a maximum pressure of 64 mm Hg. During this assessment participants were asked to report when they had the first sensation. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: 1 hour after drug was ingested
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
mm Hg | 42.83 (12.73) | 40.33 (17.17) | 44.44 (13.05)

4. Secondary Outcome: Post-Treatment Overall Sensory Rating in Response to 16, 24, 32, and 40 mm Hg Distensions
Description: The sensory rating was measured by a 100 mm long Visual Analog Scale (VAS). The VAS does not have any pre-set marks between the extremes of 0 for no pain and 100 mm for extreme pain. The investigator measures the mark made by the participant in mm and records this for the value of pain.
Time Frame: 1 hour after drug was ingested
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: mm
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
mm
  16 mm Hg Distension | 38.18 (4.68) | 38.71 (4.64) | 37.0 (4.57)
  24 mm Hg Distension | 49.64 (5.83) | 42.75 (5.16) | 39.76 (5.06)
  32 mm Hg Distension | 58.36 (5.14) | 45.35 (4.83) | 46.76 (4.78)
  40 mm Hg Distension | 57.18 (5.42) | 48.17 (4.97) | 45.52 (4.44)

5. Secondary Outcome: Fasting Colonic Tone
Description: as for outcome 2
Time Frame: After 12 hour fast, before drug administered
Population: Intention-to-treat analysis
Measure: Mean (Standard Error); unit: mL
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 24
mL | 117.8 (7.97) | 118.5 (6.41) | 114.3 (5.50)

6. Secondary Outcome: Postprandial Colonic Motility Index
Description: Colonic phasic pressure activity is summarized as a motility index (MI)=log_e[number of contractions * sum of amplitudes) + 1]. A normal fasting average motility index (MI) would be about 12. An increase in MI means an increase in the phasic contractions (in contrast to tone) which is measured as a change in volume of the barostat balloon. (Therefore, an increase in MI means that the meal is moving more quickly through the colon.)
Time Frame: 1 hour after ingestion of standard meal
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: log mm Hg
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
log mm Hg
  Proximal descending colon | 11.24 (1.13) | 11.22 (1.56) | 10.70 (2.51)
  Distal descending colon | 9.97 (2.8) | 10.23 (1.92) | 10.50 (1.69)

7. Secondary Outcome: Post-treatment Sensory Threshold for First Sensation
Description: The sensory threshold for first sensation was measured by stepwise inflation in increments of 4 mm Hg at 60 second intervals up to a maximum pressure of 64 mm Hg. During this assessment participants were asked to report when they had the first sensation. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: 1 hour after drug was ingested
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
mm Hg | 15.83 (9.62) | 15.5 (11.46) | 18.37 (14.65)

8. Secondary Outcome: Post-Treatment Sensory Threshold for First Perception of Gas
Description: The sensory threshold for first perception of gas was measured by stepwise inflation in increments of 4 mm Hg at 60 second intervals up to a maximum pressure of 64 mm Hg. During this assessment participants were asked to report when they had the first sensation. The investigator recorded the threshold pressure at which the participants reported this sensation.
Time Frame: 1 hour after drug was ingested
Population: Intention-to-treat analysis
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Number analyzed (Participants) | 24 | 24 | 27
mm Hg | 28.83 (17.57) | 27.33 (17.36) | 29.04 (16.81)

ADVERSE EVENTS:
Arm/Group | Dronabinol 2.5 mg | Dronabinol 5 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/27
Other Adverse Events (participants affected / at risk) | 10/24 | 13/24 | 10/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dronabinol 2.5 mg (N=24) | Dronabinol 5 mg (N=24) | Placebo (N=27)
Drowsy/tired (General disorders) | 5 (5) | 7 (7) | 5 (5)
Flushing/hot (General disorders) | 6 (6) | 4 (4) | 4 (4)
Headache (General disorders) | 4 (4) | 2 (2) | 4 (4)
Dizzy/light-headed (General disorders) | 2 (2) | 5 (5) | 1 (1)
Loopy/foggy thinking (General disorders) | 2 (2) | 6 (6) | 0 (0)
Elevated heart rate (Cardiac disorders) | 2 (2) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No